CLINICAL TRIAL: NCT02245477
Title: Evaluation of Maternal Serum VEGF in Pregnant Women With Foetal Growth Restriction
Brief Title: Maternal Serum Vascular Endothelial Growth Factor in Pregnant Women With Foetal Growth Restriction
Acronym: VEGF in FGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Lecturer of Obstetrics and Gynecology, Beni-Suef University
Other Study IDs: Beni-Suef 5
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Foetal Growth Restriction
Keywords: Serum VEGF, FGR
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obstetric Ultrasoud: Transabdominal ultrasound was performed to confirm foetal number, viability, gestational age, exclusion of congenital anomalies, and assessment of amniotic fluid index and localization of the placenta.
  Interventions: Device: obstetric Ultrasound
- Serum Vascular Endothelial Growth Factor: Serum VEGF concentration will be determined by Enzyme Linked immunosorbant assay using Quantitative Human VEGF Immunoassay kit (cat. No. DVEOO) manufactured by R & D Systems, Inc , (Minneapolis, MN, USA).
  Interventions: Other: serum Vascular Endothelial Growth Factor

INTERVENTIONS:
Device: obstetric Ultrasound — Transabdominal ultrasound was performed to confirm foetal number, viability, gestational age, exclusion of congenital anomalies, and assessment of amniotic fluid index and localization of the placenta.
  Groups: Obstetric Ultrasoud
Other: serum Vascular Endothelial Growth Factor — Maternal blood samples (10 cc) were taken from an antecubital vein. Plastic clean sterile tubes were used for collection of blood. Two cc of the blood sample were put in other clean sterile tubes containing ethylene diamine tetra-acetic acid (EDTA) to be used in measuring maternal hemoglobin concentrations and evaluating the complete blood count. The rest of maternal blood samples were centrifuged within 3 hours and sera collected equally in 2 suitable containers and stored at -80 degrees until assayed (first container for routine laboratory investigations and the second for VEGF assay).VEGF sample was allowed to clot for 30 minutes before centrifugation for 15 minutes. Serum is removed and assay immediately or sample was stored at -80 degrees
  Groups: Serum Vascular Endothelial Growth Factor

SUMMARY:
In this study we explore To explore the role of maternal serum vascular endothelial growth factor (VEGF) in pregnancies complicated by foetal growth restriction.

DETAILED DESCRIPTION:
Small-for-gestational age (SGA) is defined as an estimated foetal weight (EFW) or abdominal circumference (AC) less than the 10th centileand severe SGA as an EFW or AC less than the 3rd centile. Foetal Growth Restriction refers to failure of the foetus to achieve its predetermined growth potential for various reasons.Foetus with foetal growth restriction (FGR) greatly contributes to perinatal mortality and short- and long-term morbidity. There is a 3-10 fold increase in perinatal mortality in pregnancies complicated by this FGR .The incidence of FGR in newborns ranges between 3 and 7% of the total population .FGR is thought to stem from placental hypoxia-induced vasoconstriction of the fetoplacental vessels, leading to placental hypoperfusion and thus fetal undernutrition. However, the effects of hypoxia on the fetoplacental vessels have been surprisingly little studied.Vascular endothelial growth factor (VEGF) is one of the factors that take part in placental angiogenesis. It is highly expressed during embryonic and foetal development..Angiogenesis involves the branching of new microvessles from pre-existing larger blood vessels.Angiogenesis plays a role in the development of the villous vasculature and the formation of terminal villi in human placenta. IUGR occurs as a result of the failure of elongation, branching and dilatation of the capillary loops and of terminal villous formation.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* Gestational age 28-36 weeks
* Fetal growth restriction
* Patient consents to the procedure.
* BMI 20-30

Exclusion Criteria:

* Preeclampsia
* Diabetes Mellitus
* Fetal congenital anomalies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with gestational age 28-36 weeks were included in our study. Patients with SGA were defined by obstetric ultrasound as estimated fetal weight was below the10thcentile.Twice weekly CTGs and Umbilical artery (UA) Doppler were done. Women with abnormal CTGs or UA Doppler were excluded from the study. A follow up scan was done 2 weeks later and FGR will be diagnosed if fetal weight had faltered.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Obstetric ultrasound | from 28 weeks gestation to 36 weeks gestation
  Patients with gestational age 28-36 weeks were included in our study. Patients with SGA were defined by obstetric ultrasound as estimated fetal weight was below the10thcentile. Twice weekly CTGs and Umbilical artery (UA) Doppler were done. Women with abnormal CTGs or UA Doppler were excluded from the study. A follow up scan was done 2 weeks later and FGR will be diagnosed if fetal weight had altered.

SECONDARY OUTCOMES:
Serum Vascular Endothelial growth factor | 3 months until delivery
  Maternal blood samples (10 cc) were taken from an antecubital vein. Plastic clean sterile tubes were used for collection of blood. Two cc of the blood sample were put in other clean sterile tubes containing ethylene diamine tetra-acetic acid (EDTA) to be used in measuring maternal hemoglobin concentrations and evaluating the complete blood count. The rest of maternal blood samples were centrifuged within 3 hours and sera collected equally in 2 suitable containers and stored at -80 degrees until assayed (first container for routine laboratory investigations and the second for VEGF assay).VEGF sample was allowed to clot for 30 minutes before centrifugation for 15 minutes. Serum is removed and assay immediately or sample was stored at -80 degrees.Serum VEGF concentration was determined by Enzyme Linked immunosorbant assay using Quantitative Human VEGF Immunoassay kit (cat. No. DVEOO) manufactured by R & D Systems, Inc , (Minneapolis, MN, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Egypt